CLINICAL TRIAL: NCT06020469
Title: Comparative Effects of Ciprofol and Propofol on Pain Intensity of the Patients Without PCA on the First Day After Surgery: a Retrospective, Propensity Score Matched, Cohort Study
Brief Title: Comparative Effects of Ciprofol and Propofol on Pain Intensity on the First Day After Surgery: a Retrospective, Propensity Score Matched, Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Hui Zhang, associate chief physician, Guangdong Second Provincial General Hospital
Other Study IDs: GD2HMZK
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia; Acute Pain; Risk Reduction
Keywords: Data Platform; Machine Learning; Postoperative Acute Pain
MeSH Terms: conditions — Acute Pain; Risk Reduction Behavior; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Numeric Rating Scale (NRS) score after surgery <4
- Numeric Rating Scale (NRS) score after surgery ≥ 4

SUMMARY:
Data intelligence platform was widely used to facilitate the process of clinical research. However, a platform that integrates natural language processing (NLP) and machine learning (ML) algorithms has not been reported in perioperative medical management.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they were above 18 years old, undergoing non-local anesthesia surgery.

Exclusion Criteria:

* The basic information such gender, age, height, weight, and body mass index (BMI) were missing.
* Patients undergoing day surgery, with a history of multiple operations, or entering ICU after surgery, and losing the NRS score during movement at 24h after surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pain assessment was used by Numeric Rating Scale (NRS) score after surgery.
Sampling Method: Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | October 2022 to October 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China